CLINICAL TRIAL: NCT01898403
Title: Testing the Efficacy of Indocyanine Green Imaging (ICG-SPY) in the Identification of Sentinel Lymph Nodes (SLN) in Patients With Malignant Melanoma
Brief Title: Lymph Node Mapping Using Indocyanine Green Solution in Diagnosing Patients With Malignant Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ralph Greco, Johnson and Johnson Professor of Surgery, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-27319; NCI-2013-01286 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MEL0010 (Other: OnCore); P30CA124435 (NIH)
Record Dates: First submitted 2013-07-03; First posted 2013-07-12 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2015-06

CONDITIONS: Recurrent Melanoma
MeSH Terms: conditions — Melanoma | interventions — Indocyanine Green; iso-sulfan blue; Lymphoscintigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sentinel Lymph Node (SLN) Detection (Experimental): All patients receive peri-tumoral, intradermal injections of isosulfan blue and indocyanine green solution for detection of melanoma in lymph nodes. In addition, lymphoscintigraphy with 99-technetium (99Tc) sulfur colloid (TSC) will be conducted for all participants with the same objective.
  Interventions: Drug: Indocyanine green solution; Drug: Isosulfan blue (ISB); Diagnostic Test: Lymphoscintigraphy with 99-technetium (99Tc) sulfur colloid (TSC)

INTERVENTIONS:
Drug: Indocyanine green solution — Administered peri-tumoral and intradermally
  Other Names: IC-GREEN (ICG); ICG solution
Drug: Isosulfan blue (ISB) — Administered peri-tumoral and intradermally
  Other Names: Lymphazurin; N-[4-[4-(diethylamino)phenyl] (2,5-disulfophenyl) Methylene]-2,5-cyclohexadien-1-ylidene]-N-ethylethanaminium hydroxide
Diagnostic Test: Lymphoscintigraphy with 99-technetium (99Tc) sulfur colloid (TSC)
  Other Names: TSC lymph node mapping

SUMMARY:
This clinical trial compares and contrasts lymph node mapping using indocyanine green (IC-GREEN), isosulfan blue (ISB), and TSC and Lymphoscintigraphy with 99-technetium (99Tc) sulfur colloid (TSC).

Study participants with malignant melanoma will undergo all 3 evaluations to assess the extent of the spread of the melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To show that indocyanine green (ICG) (indocyanine green solution) is equal to both isosulfan blue (ISB) and technetium Tc 99m sulfur colloid (TSC) and will allow all lymph node mapping to occur in the operating room (OR).

OUTLINE:

Patients receive peri-tumoral, intradermal injections of isosulfan blue and indocyanine green solution. During surgery, patients undergo identification of the sentinel lymph node and imaging using a laser with videocamera (SPY Elite camera).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign informed consent document
* Signed written informed consent
* Malignant melanoma (MM) undergoing sentinel lymph node biopsy (SNLB)
* 18 years of age or older
* Complete blood count (CBC) and metabolic panel within 6 months

Exclusion Criteria:

* History of hepatic or renal failure
* Allergy to iodine containing products
* Pregnant or may be pregnant
* Psychiatric or addictive disorders that in the opinion of the research team, may not be able to meet study requirements
* Undergoing dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Greco, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sentinel Lymph Node (SLN) Detection: All patients receive peri-tumoral, intradermal injections of isosulfan blue and indocyanine green solution for detection of melanoma in lymph nodes. In addition, lymphoscintigraphy with 99-technetium (99Tc) sulfur colloid (TSC) will be conducted for all participants with the same objective.
  Indocyanine green solution: Administered peri-tumoral and intradermally
  Isosulfan blue (ISB): Administered peri-tumoral and intradermally
  Lymphoscintigraphy with 99-technetium (99Tc) sulfur colloid (TSC)
Period: Overall Study
Arm/Group | Sentinel Lymph Node (SLN) Detection
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sentinel Lymph Node (SLN) Detection
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 31
  >=65 years | 18
Age, Continuous [Mean (Full Range); unit: years] | 60.7 [18.9 to 86.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 44
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Sentinel Lymph Nodes (SLN) Mapping
Description: Sentinel lymph nodes (SLN) will be identified and mapped using indocyanine green (ICG) solution, isosulfan blue (ISB) solution, and TSC lymphoscintigraphy.
Time Frame: Up to 1 year
Population: All participants were evaluated for sentinel lymph nodes (SLN) using Isosulfan Blue (ISB); Indocyanine Green (ICG); and TSC lymphoscintigraphy.
Measure: Number; unit: Sentinel lymph nodes
Units Other Than Participants: Sentinel Lymph Nodes
Groups:
- Sentinel Lymph Node (SLN) Detection by Isosulfan Blue; Sentinel Lymph Node (SLN) Detection by Indocyanine Green; Sentinel Lymph Node (SLN) Detection by TSC Lymphoscintigraphy: All patients received peri-tumoral, intradermal injections of isosulfan blue and indocyanine green solution for detection of melanoma in lymph nodes. In addition, lymphoscintigraphy with 99-technetium (99Tc) sulfur colloid (TSC) will be conducted for all participants with the same objective.
Arm/Group | Sentinel Lymph Node (SLN) Detection by Isosulfan Blue | Sentinel Lymph Node (SLN) Detection by Indocyanine Green | Sentinel Lymph Node (SLN) Detection by TSC Lymphoscintigraphy
Number analyzed (Participants) | 50 | 50 | 50
Number analyzed (Sentinel Lymph Nodes) | 61 | 61 | 61
Sentinel lymph nodes
  SLN detected by ISB, ICG, and TSC | 25 | 25 | 25
  SLN detected by ISB and TSC only | 4 | 0 | 4
  SLN detected by ICG and TSC only | 0 | 9 | 9
  SLN detected by ISB and ICG only | 10 | 10 | 0
  SLN detected by ISB plus any/none | 41 | 0 | 0
  SLN detected by ISB only | 2 | 0 | 0
  SLN detected by ICG plus any/none | 0 | 47 | 0
  SLN detected by ICG only | 0 | 3 | 0
  SLN detected by TSC plus any/none | 0 | 0 | 41
  SLN detected by TSC only | 0 | 0 | 3

ADVERSE EVENTS:
Arm/Group | Sentinel Lymph Node (SLN) Detection
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 5/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sentinel Lymph Node (SLN) Detection (N=50)
Infection (Infections and infestations) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No